CLINICAL TRIAL: NCT00158353
Title: Development and Evaluation of a Youth Mentoring Program
Brief Title: Evaluation of a Youth Mentoring Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Big Brothers Big Sisters of Metropolitan Chicago (Unknown)
Responsible Party: Principal Investigator, David DuBois, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003-0689; R21MH069564 (NIH); DSIR 84-CTP
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Self Concept
Keywords: Mentors; Self-esteem; Adolescent; Mental health; Social support; Substance use; Violence; Exercise; Nutrition; Sexual behavior; Female
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Motor Activity; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GirlPOWER! mentoring program
  Interventions: Behavioral: GirlPOWER! mentoring program
- 2 (Active Comparator): Big Brothers Big Sisters community-based mentoring program
  Interventions: Behavioral: Traditional mentoring

INTERVENTIONS:
Behavioral: GirlPOWER! mentoring program — GirlPOWER! mentoring program includes monthly 3-hour workshops for youth and mentors combined with monthly supplemental activities to be completed independently by youth-mentor pairs.
  Arms: 1
Behavioral: Traditional mentoring — Traditional mentoring includes a community-based mentoring program, in which the youth-mentor spends time together in activities of their choosing 2 to 4 times a month.
  Other Names: Big Brothers Big Sisters Community-Based Mentoring Program
  Arms: 2

SUMMARY:
This study will be used to determine the effectiveness of GirlPOWER!, an innovative mentoring program for adolescent minority girls living in urban areas.

DETAILED DESCRIPTION:
The potential benefits of adolescent mentoring programs cannot be overemphasized. Mentoring may be especially beneficial to urban-living, minority adolescents who may lack role models. The Big Brothers Big Sisters (BBBS) organization administers a widely-praised and empirically-supported program that is committed to building successful mentoring relationships between adolescents and adults in their community. In collaboration with the BBBS affiliate agency in Chicago, the PI has developed an intervention called GirlPOWER! GirlPOWER! combines mentoring with self-esteem enhancement and health education and promotion strategies. This study will determine the effectiveness of the GirlPOWER! intervention and determine its feasibility in being applied to other populations.

Participants will be randomly assigned to receive either the GirlPOWER! intervention or traditional mentoring through BBBS and followed for 1 year. Participants in the GirlPOWER! group and their mentors will engage in structured activities that focus on strengthening the mentoring relationship, promoting self-esteem, reducing levels of health-compromising behaviors such as substance use and violence, and increasing levels of health-enhancing behaviors. Traditional mentoring comprises less structured activities and typically includes general discussion of an adolescent's day-to-day life and any accomplishments and challenges he or she may have experienced. Participants will be assessed at study entry, 3 months following entry, and at the end of one year. Assessments will include surveys completed by youth as well as their parents, mentors, and teachers; academic data also will be obtained from school records.

ELIGIBILITY:
Inclusion Criteria:

* Live in Chicago, Illinois Metropolitan area
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

-Significant cognitive limitations or behavioral concerns that would preclude ability to participate appropriately in the intervention

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
Mental health | Measured at Year 1
  Composite measure that is the average of T-scores for Internalizing and Externalizing scales of the Youth Self-Report and Child Behavior Checklist of the Achenbach System of Empirically-Based Assessment
Health behaviors | Measured at Year 1
  Composite (average) of standardized (M=0, SD=1) scores on measures of exercise (3 items), healthy eating (10 items), unhealthy weight loss behaviors (reverse-weighted) (3 items) and substance use (reverse-weighted) (5 items) from the CDC Youth Risk Behavior Surveillance System

SECONDARY OUTCOMES:
Social support | Measured at Year 1
  Composite (average) of Friend, Family, and Very Important Adults subscales of the Perceived Support Scale-Revised, with Very Important Adults scored 0 for those reporting no very important adults.
Academic achievement | Measured at Year 1
  Composite of averages of grades reported in core subject area classes (Language Arts, Math,Science, Social Studies) by youth and parent

CONTACTS AND LOCATIONS:
Overall Officials: David L. DuBois, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] DuBois DL, Holloway BE, Valentine JC, Cooper H. Effectiveness of mentoring programs for youth: a meta-analytic review. Am J Community Psychol. 2002 Apr;30(2):157-97. doi: 10.1023/A:1014628810714. PMID 12002242
- [Background] DuBois, D. L., Silverthorn, N., Pryce, J., Reeves, E., Sanchez, B., Silva, A., Ansu, A. A., Haqq, S., & Takehara, J. (in press). Mentorship: The GirlPOWER! program. To appear in C. W. Leroy & J. E. Mann (Eds.), Handbook of preventive and intervention programs for adolescent girls. Hoboken, NJ: Wiley.
- [Background] Keller TE, Overton B, Pryce JM, Barry JE, Sutherland A, DuBois DL. "I really wanted her to have a Big Sister": Caregiver perspectives on mentoring for early adolescent girls. Child Youth Serv Rev. 2018 May;88:308-315. doi: 10.1016/j.childyouth.2018.03.029. Epub 2018 Mar 19. PMID 30323545
- [Result] Sanchez B, Pryce J, Silverthorn N, Deane KL, DuBois DL. Do mentor support for ethnic-racial identity and mentee cultural mistrust matter for girls of color? A preliminary investigation. Cultur Divers Ethnic Minor Psychol. 2019 Oct;25(4):505-514. doi: 10.1037/cdp0000213. Epub 2018 Oct 1. PMID 30272473
- [Result] Pryce JM, Silverthorn N, Sanchez B, DuBois DL. GirlPOWER! Strengthening mentoring relationships through a structured, gender-specific program. New Dir Youth Dev. 2010 Summer;2010(126):89-105. doi: 10.1002/yd.351. PMID 20665833
- See also: MENTOR/National Mentoring Partnership — http://mentoring.org
- See also: Big Brothers Big Sisters of Metropolitan Chicago — http://www.bbbschgo.org/